CLINICAL TRIAL: NCT05272514
Title: Impact of Hypoxia on Resting and Exertional Right Ventricular Performance - A PILOT STUDY
Brief Title: Impact of Hypoxia on Resting and Exertional Right Ventricular Performance
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 21-4354
Record Dates: First submitted 2022-02-08; First posted 2022-03-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Ventricular Dysfunction, Right; Hypoxia
MeSH Terms: conditions — Ventricular Dysfunction, Right; Hypoxia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy individuals: 10 healthy individuals will be recruited.
  Interventions: Other: Hypoxia

INTERVENTIONS:
Other: Hypoxia — Individuals will be exposed to varying levels of hypoxia according to the protocol detailed above.

SUMMARY:
The purpose of this study is to better understand how hypoxia (low oxygen) affects resting and exertional right ventricular function in healthy individuals.

DETAILED DESCRIPTION:
The right ventricle plays a critical role in exercise. As workload increases with exercise, the right ventricle augments contractility and lusitropy (diastolic relaxation) to accommodate increased venous return (preload) and pulmonary arterial pressure (afterload). Using gold-standard pressure-volume analysis, the investigators have shown that impairments in right ventricular function limit functional capacity among individuals with cardiovascular disease, heart failure and pulmonary hypertension. In addition, the investigators have characterized right ventricular function during exercise in the healthy heart using these techniques. Hypoxia increases pulmonary arterial pressure via hypoxic pulmonary vasoconstriction. By increasing right ventricular afterload, hypoxia may compromise exercise capacity. However, data regarding the impact of hypoxia on right ventricular performance are lacking.

This is a human physiology study of resting and exertional right ventricular function under control (normoxic) and hypoxic conditions. The investigators will use pressure-volume analysis in conjunction with Swan-Ganz catheterization and echocardiography to assess right ventricular performance in healthy individuals at rest and during exercise in normoxia and hypoxia. The study protocol consists of three visits.

* Visit 1: Non-invasive symptom-limited cardiopulmonary exercise test under normoxic conditions (FiO2= 0.21).
* Visit 2: Non-invasive symptom-limited cardiopulmonary exercise test under hypoxic conditions (FiO2=0.12).
* Visit 3: Invasive resting and exertional hemodynamic assessment under normoxic and hypoxic conditions

In Visits 1 and 2, heart rate/rhythm, oxygen saturation, blood pressure, gas exchange parameters (oxygen uptake [VO2], carbon dioxide production [VCO2], and minute ventilation), and rated perceived exertion will be monitored. Cardiopulmonary exercise testing (CPET) will be performed on an upright cycle ergometer with workload starting at 0 Watts and increasing every 2 minutes until volitional exhaustion with maximum workload at 8-12 minutes. The order of Visits 1 and 2 will be randomized to reduce the potential for bias from a learning/ordering effect.

In Visit 3, the same non-invasive measurements will be obtained. Additionally, right heart catheterization with Swan-Ganz catheter and conductance catheter placement will be performed. This will provide gold-standard hemodynamic and pressure-volume loop analysis to measure outcomes of right ventricular contractility, lusitropy (diastolic relaxation), afterload, and ventricular-arterial coupling. First, participants will complete submaximal exercise at FiO2=0.21. Submaximal exercise will include 5 minutes at 50% of baseline maximal oxygen uptake (VO2max achieved during Visit 1). After 20 minutes' rest, hemodynamic measurements will be obtained at rest at FiO2 0.21, 0.17, 0.15 and 0.12 to characterize the impact of progressive hypoxia on resting right ventricular hemodynamics. Participants will then perform submaximal exercise (50% VO2 max from hypoxic baseline at Visit 2) at FiO2 0.12. Thereafter, participants will complete a symptom-limited CPET at FiO2 0.12 with monitoring of invasive hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 60
* For women, premenopausal status

Exclusion Criteria:

* Active cardiovascular or pulmonary disease (e.g. hypertension, coronary artery disease, cardiomyopathy, arrhythmia, valvular abnormalities, diabetes, peripheral vascular disease, tobacco use, chronic obstructive pulmonary disease, asthma, interstitial lung disease, restrictive lung disease, or pulmonary hypertension)
* Use of cardiac- or pulmonary-related medications
* Prior history of high altitude pulmonary edema or high altitude cerebral edema
* Body mass index < 18.5 or > 30
* Anemia
* Iron deficiency
* Iron supplementation (oral or intravenous) in the preceding 60 days
* Systemic anticoagulation or aspirin use that cannot be temporarily held for the study
* Pregnancy
* Non-cardiopulmonary disorders that adversely influence exercise ability (e.g. arthritis or peripheral vascular disease)
* Dedicated athletic training (defined here as spending >9 hours per week in vigorous physical activity [≥6 mets])
* Regular high-altitude exercise (defined here as engaging in vigorous physical activity [≥1 hour at ≥6 mets] at ≥8,000 ft for >2 days per week over the preceding 4 weeks)
* Residence at ≥8,000 ft for 3 or more consecutive nights in the preceding 30 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 10 healthy men and women
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Right ventricular contractility measured by conductance catheter | Up to 1 hour
  End-systolic elastance (Ees) in mmHg/mL
Right ventricular lusitropy (diastolic function) measured by conductance catheter | Up to 1 hour
  Minimum dp/dt in mmHg/sec

SECONDARY OUTCOMES:
Right ventricular stroke work measured by conductance catheter | Up to 1 hour
  Area of pressure-volume loop
Mean pulmonary artery pressure measured by right heart catheterization | Up to 1 hour
  In mmHg
Cardiac output derived from right heart catheterization | Up to 1 hour
  In L/min, calculated by Fick equation
Workload | Up to 1 hour
  Workloads attained with submaximal and maximal exercise testing
Maximal oxygen uptake | Up to 1 hour
  VO2max achieved in maximal exercise testing
Plasma acylcarnitine 10:0 measured by peripheral venous metabolomics (ultra-high performance liquid chromatography coupled to mass spectrometry) | Up to 1 hour
  Relative ion count
Red blood cell acylcarnitine 10:0 measured by peripheral venous metabolomics (ultra-high performance liquid chromatography coupled to mass spectrometry) | Up to 1 hour
  Relative ion count

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith TG, Balanos GM, Croft QP, Talbot NP, Dorrington KL, Ratcliffe PJ, Robbins PA. The increase in pulmonary arterial pressure caused by hypoxia depends on iron status. J Physiol. 2008 Dec 15;586(24):5999-6005. doi: 10.1113/jphysiol.2008.160960. Epub 2008 Oct 27. PMID 18955380
- [Background] Smith TG, Talbot NP, Privat C, Rivera-Ch M, Nickol AH, Ratcliffe PJ, Dorrington KL, Leon-Velarde F, Robbins PA. Effects of iron supplementation and depletion on hypoxic pulmonary hypertension: two randomized controlled trials. JAMA. 2009 Oct 7;302(13):1444-50. doi: 10.1001/jama.2009.1404. PMID 19809026
- [Background] Cornwell WK, Tran T, Cerbin L, Coe G, Muralidhar A, Hunter K, Altman N, Ambardekar AV, Tompkins C, Zipse M, Schulte M, O'Gean K, Ostertag M, Hoffman J, Pal JD, Lawley JS, Levine BD, Wolfel E, Kohrt WM, Buttrick P. New insights into resting and exertional right ventricular performance in the healthy heart through real-time pressure-volume analysis. J Physiol. 2020 Jul;598(13):2575-2587. doi: 10.1113/JP279759. Epub 2020 May 18. PMID 32347547
- [Background] Cornwell WK 3rd, Baggish AL, Bhatta YKD, Brosnan MJ, Dehnert C, Guseh JS, Hammer D, Levine BD, Parati G, Wolfel EE; American Heart Association Exercise, Cardiac Rehabilitation, and Secondary Prevention Committee of the Council on Clinical Cardiology; and Council on Arteriosclerosis, Thrombosis and Vascular Biology. Clinical Implications for Exercise at Altitude Among Individuals With Cardiovascular Disease: A Scientific Statement From the American Heart Association. J Am Heart Assoc. 2021 Oct 5;10(19):e023225. doi: 10.1161/JAHA.121.023225. Epub 2021 Sep 9. PMID 34496612
- [Derived] Forbes LM, Bull TM, Lahm T, Lawley JS, Hunter K, Levine BD, Lovering A, Roach RC, Subudhi AW, Cornwell WK 3rd. Right Ventricular Response to Acute Hypoxia among Healthy Humans. Am J Respir Crit Care Med. 2023 Aug 1;208(3):333-336. doi: 10.1164/rccm.202303-0599LE. No abstract available. PMID 37311248